CLINICAL TRIAL: NCT03453892
Title: Investigation of the Timely-coordinated Therapy of Patients With Metastatic Cancer by Radiotherapy Together With Immune Checkpoint Inhibition
Acronym: ST-ICI
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: ST-ICI
Record Dates: First submitted 2018-01-24; First posted 2018-03-05 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Cancer
Keywords: Metastatic cancer; Radiotherapy; Immunotherapy; radioimmuno therapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Nivolumab; pembrolizumab; Radiotherapy; Ipilimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Blood cells, circulating DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anti CTLA-4: The study cohort consist of patients suffering from metastatic cancer of several entities which will be treated with palliative RT and/or ICI (anti CTLA-4) at Department of Radiation Oncology of Universitätsklinikum Erlangen.
  Interventions: Radiation: Radiotherapy; Drug: Ipilimumab
- anti PD-1/PD-L1: The study cohort consist of patients suffering from metastatic cancer of several entities which will be treated with palliative RT and/or ICI (anti PD-1/PD-L1) at Department of Radiation Oncology of Universitätsklinikum Erlangen.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nivolumab — The normal clinical treatment-plan of the underlying disease remains unchanged.
  Groups: anti PD-1/PD-L1
Drug: Pembrolizumab — The normal clinical treatment-plan of the underlying disease remains unchanged.
  Groups: anti PD-1/PD-L1
Radiation: Radiotherapy — The normal clinical treatment-plan of the underlying disease remains unchanged.
Drug: Ipilimumab — The normal clinical treatment-plan of the underlying disease remains unchanged.
  Groups: anti CTLA-4

SUMMARY:
Immunotherapy for the treatment of several cancer entities steadily increased during the last years. The data from the finalized and ongoing studies show the tremendous impact of immune checkpoint inhibition (ICI) also for advanced metastatic patients. Especially the ICI with pembrolizumab and nivolumab have an increasing number of first line treatment approvals. However, in particular metastatic patients which receive ICI therapy are often irradiated for immediate palliation of several metastases. Preclinical work revealed that radiotherapy (RT) is capable to modulate the tumor phenotype, its microenvironment in a way that systemic anti-tumor immune responses are induced. However, radiation has also immune suppressive properties as e.g. the expression of immune checkpoint molecules is increased following radiotherapy. So the ICI therapy in combination with the RT has the potential to overcome the immunotolerance of the tumor and the metastases. More and more reports therefore describe a so-called systemic immune-modulating effect of radiotherapy (former and still often named as abscopal effect). However the timely application of ICI and RT is often randomly and depends on the clinical need for the palliative RT. The aim of this trial is therefore to standardize the chronology of RT in combination with ICI, to evaluate the effects of radio-immunotherapy with a stratified and comparable patient cohort. The ST-ICI study is a prospective and observational study not influencing the standard therapeutic scheme and will provide hints how the radio-immune therapy drives systemic anti tumor responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering and diagnosed for: metastatic cancer of several entities
* Clinical indicated therapy with PD-1/PD-L1 inhibitors or CTLA-4 antagonists
* Optionally radiotherapy if clinically indicated
* Age at least 18 years

Exclusion Criteria:

* fertile patients who refuse effective contraception during study treatment
* persistent drug and/or alcohol abuse
* patients not able or willing to behave according to study protocol
* patients in care
* patients that are not able to speak German
* patients which are imprisoned according to legal or governmental order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort consist of patients suffering from metastatic cancer of several entities which will be treated with optionally RT (if indicated) and/or ICI at Department of Radiation Oncology of Universitätsklinikum Erlangen.
  Both gender are included into the study, a maximum age was not defined.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Systemic (according to iRECIST criteria) and local response of detected metastases during radio and/or immunotherapy. | From date of inclusion to the trial until the date of first documented iRECIST progression or date of death from any cause, whichever came first, assessed up to day 540.
Change of circulating immune cells of treated patients by deep immunophenotyping. | The analyses are conducted at time points before (day 0) and before every prescription of ICI (every 14 to 21 days) till progression or end of study at day 540
  Immunophenotyping of the patients: Detection of about 30 distinct immune sell (sub)types together with their activation markers. The analyses are conducted at time points before (day 0) and before every prescription of ICI (every 14 to 21 days) till progression or end of study at day 540.

SECONDARY OUTCOMES:
Detection of adverse events according to NCI CTAE (v4.0) | From date of inclusion to the trial until the date of first documented iRECIST progression or date of death from any cause, whichever came first, assessed up to day 540.
Documentation of corticoid prescription | From date of inclusion to the trial until the date of first documented iRECIST progression or date of death from any cause, whichever came first, assessed up to day 540.
Overall survival | Till death of the patient or end of study at day 540, whichever came first
Progression free survival | From date of inclusion to the trial until the date of first documented iRECIST progression or date of death from any cause, whichever came first, assessed up to day 540.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, Prof. Dr., Study Chair — Department of Radiation Oncology, Universitätsklinikum Erlangen; Markus Hecht, Dr. med., Study Director — Department of Radiation Oncology, Universitätsklinikum Erlangen; Udo S Gaipl, Prof. Dr., Study Director — Department of Radiation Oncology, Universitätsklinikum Erlangen
Locations (1):
- Department of Radiation Oncology, Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Griewing LM, Schweizer C, Schubert P, Rutzner S, Eckstein M, Frey B, Haderlein M, Weissmann T, Semrau S, Gostian AO, Muller SK, Traxdorf M, Iro H, Zhou JG, Gaipl US, Fietkau R, Hecht M. Questionnaire-based detection of immune-related adverse events in cancer patients treated with PD-1/PD-L1 immune checkpoint inhibitors. BMC Cancer. 2021 Mar 24;21(1):314. doi: 10.1186/s12885-021-08006-0. PMID 33761922
- [Derived] Zhou JG, Donaubauer AJ, Frey B, Becker I, Rutzner S, Eckstein M, Sun R, Ma H, Schubert P, Schweizer C, Fietkau R, Deutsch E, Gaipl U, Hecht M. Prospective development and validation of a liquid immune profile-based signature (LIPS) to predict response of patients with recurrent/metastatic cancer to immune checkpoint inhibitors. J Immunother Cancer. 2021 Feb;9(2):e001845. doi: 10.1136/jitc-2020-001845. PMID 33593828